CLINICAL TRIAL: NCT01676675
Title: A Single Center, Randomized, Double-blind, Placebo-controlled, Dose-escalation Phase I Clinical Trial for Safety and Preliminary Immunogenicity of a Whole Virus Inactivated Influenza H5N1 Vaccine in Healthy Adolescents and Adults, on Day 0 and 21 Intramuscularly
Brief Title: A Phase I Clinical Trial With Whole Virus Inactivated Influenza H5N1 Vaccine in Healthy Adolescents and Adults
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Wuhan Institute of Biological Products Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT011
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: whole virus; inactivated; influenza; H5N1 vaccine; safety; immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 7.5μg/0.5ml in subjects(12-17 years old) (Experimental): whole virus inactivated influenza H5N1 vaccine of 7.5μg /0.5ml in 30 adolescents aged 12-17 years old on day 0, 21
  Interventions: Biological: 7.5μg /0.5ml
- 15μg/0.5ml in subjects(12-17 years old) (Experimental): whole virus inactivated influenza H5N1 vaccine of 15.0μg /0.5ml in 30 adolescents aged 12-17 years old on day0,21
  Interventions: Biological: 15.0μg /0.5ml
- 30μg/0.5ml in subjects(12-17 years old) (Experimental): whole virus inactivated influenza H5N1 vaccine of 30.0μg /0.5ml in 30 adolescents aged 12-17 years old on day0,21
  Interventions: Biological: 30.0μg /0.5ml
- 7.5μg/0.5ml in subjects(18-60 years old) (Experimental): whole virus inactivated influenza H5N1 vaccine of 7.5μg /0.5ml in 30 adults aged 18-60 years old on day 0, 21
  Interventions: Biological: 7.5μg /0.5ml
- 15μg/0.5ml in subjects(18-60 years old) (Experimental): whole virus inactivated influenza H5N1 vaccine of 15.0μg /0.5ml in 30 adults aged 18-60 years old on day 0, 21
  Interventions: Biological: 15.0μg /0.5ml
- 30μg/0.5ml in subjects(18-60 years old) (Experimental): whole virus inactivated influenza H5N1 vaccine of 30.0μg /0.5ml in 30 adults aged 18-60 years old on day 0, 21
  Interventions: Biological: 30.0μg /0.5ml
- 0/0.5ml in adolescents (12-17 years old) (Placebo Comparator): 0/0.5ml placebo in 30 adolescents aged 12-17 years old on day 0, 21
  Interventions: Biological: 0/0.5ml placebo
- 0/0.5ml in adults(18-60 years old) (Placebo Comparator): 0/0.5ml placebo in 30 adults aged 18-60 years old on day 0, 21
  Interventions: Biological: 0/0.5ml placebo

INTERVENTIONS:
Biological: 7.5μg /0.5ml — whole virus inactivated influenza H5N1 vaccine of 7.5μg /0.5ml, two doses, 21 days interval
  Arms: 7.5μg/0.5ml in subjects(12-17 years old); 7.5μg/0.5ml in subjects(18-60 years old)
Biological: 15.0μg /0.5ml — whole virus inactivated influenza H5N1 vaccine of 15.0μg /0.5ml, two doses, 21 days interval
  Arms: 15μg/0.5ml in subjects(12-17 years old); 15μg/0.5ml in subjects(18-60 years old)
Biological: 30.0μg /0.5ml — whole virus inactivated influenza H5N1 vaccine of 30.0μg /0.5ml, two doses, 21 days interval
  Arms: 30μg/0.5ml in subjects(12-17 years old); 30μg/0.5ml in subjects(18-60 years old)
Biological: 0/0.5ml placebo — 0/0.5ml placebo, two doses, 21 days interval
  Arms: 0/0.5ml in adolescents (12-17 years old); 0/0.5ml in adults(18-60 years old)

SUMMARY:
Influenza is an acute respiratory infection caused by influenza virus with high incidence and serious complications even causing death. According to the announcement released by the World Health Organization (WHO), the number of global annual influenza case was 0.6 to 1.2 billion and 0.5 to 1 million people died. The emergence of a new subtype of influenza virus may cause an influenza pandemic with occurence once every 10 to 50 years which cause serious adverse consequences for human health and social welfare worldwide.

From 1997 to 2003，the H5N1 virus infection has increased highly and gradually spreaded to Europe, Africa and other countries and regions. High mortality caused by H5N1 virus has attracted the WHO and national government great attention. So it is meaningful to develop vaccine to provide effective antibody to reduce the number of infections.

The objective of this study is to evaluate the safety and preliminary immunogenicity of a whole virus inactivated influenza H5N1 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged from 12 to 60 years old of normal intelligence;
* The subjects' guardians are able to understand and sign the informed consent;
* Subjects established as healthy after medical history questioning, physical examination and clinical decision;
* Subjects who can comply with the requirements of the clinical trial protocol;
* Subjects who have never received influenza H5N1 vaccine and other preventive products;
* Subjects with temperature ≤37°C on axillary setting.

Exclusion Criteria:

Exclusion Criteria for the first dose:

* Women in pregnancy / lactation or plan to be pregnant during the study;
* The subject has a history of allergy or is allergic with any Ingredient of vaccine, such as egg, ovalbumin;
* Had serious adverse reactions in previous vaccination, such as allergies, hives, difficult breath, angioneurotic edema or abdominal pain;
* Autoimmune diseases or immune deficiency;
* Had asthma, over the past two years, the condition is unstable in need of emergency treatment, hospitalization and oral or intravenous corticosteroids;
* Diabete (type I or type II) not including gestational diabete;
* Thyroidectomy history, or treatment because of thyroid diseases in the past 12 months;
* Over the past 3 years, severe angioneurotic edema, or need treatment in the past 2 years;
* Severe hypertension and blood pressure is still more than 150/100 mmHg after drug maintenance therapy;
* coagulation abnormalities diagnosed by doctor (such as lack of coagulation factors, coagulation disorder diseases, platelet abnormality) or coagulation disorder;
* Malignancy, active or treated tumor without explicitly been cured, or the possibility of a recurrence during the study period;
* Epilepsy not including alcohol epilepsy of stop drinking in the first 3 years or the simplicity not requiring treatment in the past 3 years;
* Asplenia, functional asplenia, and any circumstances leading to asplenia or splenectomy;
* Guillain-Barre syndrome;
* Had immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding corticosteroid spray to treat allergic rhinitis and corticosteroid treatment of the acute uncomplicated dermatitis) within the past six months;
* Received immune globulin in three months before study;
* Received other experimental drugs in 30 days before study;
* Received live attenuated vaccine in 30 days before study;
* Receiving subunit or inactivated vaccines in 14days before study, such as pneumococcal vaccine or allergy treatment;
* In prevention or treatment of the anti-TB (antituberculosis) now;
* Had fever (axillary temperature ≥ 38.0℃) 3 days before vaccination or had any acute illness in the past five days requiring systemic antibiotics or antiviral therapy);
* The subject is unable to comply with the study requirements because of psychology, or had mental illness or dual-stage affective psychosis not well controlled within the past two years or had psychology in medication and suicidal tendency in the past five years;
* According to the researcher, contrary to the study protocol or effect signed informed consent due to a variety of medical, psychological, social conditions, occupational factors or other conditions.

Exclusion Criteria for the second dose:

* Had any vaccination-related Grade 3 or more adverse reactions in 72 hours after first vaccination;
* Any situation meets the exclusion criteria stated in the exclusion criteria for first dose;
* Had serious adverse reactions caused by the study vaccination.
* Acute infection;
* Any condition the investigator believed may affect the evaluation of the vaccine.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
the safety of whole virus inactivated influenza H5N1 vaccine in healthy adolescents aged from 12-17 years and adults aged from 18-60 years | 21 days after the first dose
  Frequency of systemic and local adverse reactions within 21 days after the first doses of whole virus inactivated influenza H5N1 vaccine in healthy adolescents aged from 12-17 years and adults aged from 18-60 years
the safety of whole virus inactivated influenza H5N1 vaccine in healthy adolescents aged from 12-17 years and adults aged from 18-60 years | 21 days after the second dose
  Frequency of systemic and local adverse reactions within 21 days after the second doses of whole virus inactivated influenza H5N1 vaccine in healthy adolescents aged from 12-17 years and adults aged from 18-60 years
the immunogenicity of the vaccine after first dose | on day 21±3 days
  the seroconversion rate and GMFI of antibodies on day 21 after first dose with different formulation vaccines in healthy adolescents aged from 12-17 years and adults aged from 18-60 years
the immunogenicity of the vaccine after second dose | on day 42±7 days
  the seroconversion rate and GMFI of antibodies on day 21 after second dose with different formulation vaccines in healthy adolescents aged from 12-17 years and adults aged from 18-60 years
the immunogenicity of the vaccine after whole immunization | 3 months after second dose (±14 days)
  the seroconversion rate and GMFI of antibodies 3 months after the second dose with different formulation vaccines in healthy adolescents aged from 12-17 years and adults aged from 18-60 years

SECONDARY OUTCOMES:
abnormal change of hematological examination and the function of liver and kidney after first dose | 3 days after first dose
  abnormal change of hematological examination and the function of liver and kidney 3 days after first dose with different formulation vaccines in healthy adolescents aged from 12-17 years and adults aged from 18-60 years
abnormal change of hematological examination and the function of liver and kidney after second dose | 3 days after second dose
  abnormal change of hematological examination and the function of liver and kidney 3 days after second dose with different formulation vaccines in healthy adolescents aged from 12-17 years and adults aged from 18-60 years

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China